CLINICAL TRIAL: NCT05757466
Title: Efficacy and Safety Study of Second-Line Prolgolimab Monotherapy or in Combination With Bendamustine for Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Prolgolimab Monotherapy or in Combination With Bendamustine for r/r Classical Hodgkin Lymphoma
Acronym: Prolgo-HL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Collaborators: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science RM Gorbacheva Institute, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27/22-н
Record Dates: First submitted 2023-02-17; First posted 2023-03-07 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; Prolgolimab; PD-1 inhibitors; Bendamustine; Immunotherapy; Relapsed/refractory; Autologous stem cell transplantation,
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm (Experimental): Patients receive 6 cycles of prolgolimab monotherapy with subsequent assessment of response by PET/CT using Lugano and LYRIC criteria. Patients with complete response continue prolgolimab therapy for up to 24 cycles. Patients are switched to combination therapy with prolgolimab and chemotherapy (bendamustine) if the complete response is not achieved after 6 cycles of therapy or in case of relapse during prolgolimab monotherapy.
  Patients without complete response after 6 cycles of prolgolimab monotherapy or with relapse during monotherapy will receive 3 cycles of combination therapy with prolgolimab and bendamustine every 28 days. Collection of hematopoietic stem cells is performed at any stage of combination therapy. Response evaluation after 3 cycles of combination therapy is performed by PET/CT using Lugano and LYRIC criteria. Autologous stem cell transplantation is conducted in patients who achieve complete or partial response.
  Interventions: Drug: Prolgolimab; Drug: Combination with prolgolimab and bendamustine

INTERVENTIONS:
Drug: Prolgolimab — Prolgolimab monotherapy 1 mg/kg IV every 2 weeks up to a maximum of 24 cycles
Drug: Combination with prolgolimab and bendamustine — Prolgolimab 1 mg/kg IV D1,15; Bendamustine 90 mg/m2 IV D1,2, 28-day cycle, maximum of 3 cycles;

SUMMARY:
Prolgolimab is an anti-PD-1 inhibitor that has previously been shown to be effective and safe for the treatment of patients with melanoma. Given the mechanism of action, it is expected to be effective in patients with classical Hodgkin lymphoma (cHL).

The use of PD-1 inhibitors in 2nd line treatment, as part of PET-adapted monotherapy/combination therapy, has already demonstrated a favorable toxicity profile, as well as a high efficacy, which may lead to increased survival of patients with r/r cHL. It has been demonstrated that long-term disease remission can be achieved after PD-1 inhibitor therapy, even in a group of heavily pretreated patients with relapsed/refractory cHL. The use of prolgolimab as part of PET-adapted therapy strategy in this study may allow to achieve a prolonged remission in patients with cHL who are highly sensitive to immunotherapy while omitting the autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically verified diagnosis of cHL, refractory or relapsed after the first line of therapy
* Age 18-70 y
* Ejection fraction not less than 50%
* No severe concurrent illness
* 0-2 ECOG status
* Use of highly effective contraceptive methods from the moment of signing the informed consent form, throughout the study and within 6 months after receiving the last dose of the drug.

Exclusion Criteria:

* Severe organ failure: creatinine > 2 norms; alanine aminotransferase, aspartate aminotransferase > 5 norms; bilirubin> 1.5 norms;
* Respiratory failure > grade 1 at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Active or prior documented autoimmune disease requiring systemic treatment
* Pregnancy, breastfeeding, planning pregnancy or parenthood during the study period
* Hypersensitivity or allergy to study drugs
* Somatic or mental pathology that does not allow to perform research procedures, including the signing of informed consent
* Simultaneous use of drugs or medical devices studied in other clinical trials
* Use of PD-1 inhibitors or bendamustine in the 1st line of therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate during prolgolimab monotherapy | 12 months
  Overall response rate (ORR), defined as the proportion of patients with complete response (CR) or partial response (PR) in measurable lesions as defined by Lugano and LYRIC criteria

SECONDARY OUTCOMES:
Frequency of grade 3 or higher treatment-related adverse events during prolgolimab monotherapy | 12 months
  Toxicity was graded according to NCI CTCAE 5.0.(Common Terminology Criteria for Adverse Events Version 5.0)
Frequency of grade 3 or higher treatment-related adverse events during combination therapy (prolgolimab+bendamustine) | 24 months
  Toxicity was graded according to NCI CTCAE 5.0.(Common Terminology Criteria for Adverse Events Version 5.0)
Overall response rate during combination therapy (prolgolimab+bendamustine) | 24 months
  Overall response rate (ORR), defined as the proportion of patients with complete response (CR) or partial response (PR) in measurable lesions as defined by Lugano and LYRIC criteria
1-year and 2-year overall survival | 24 months
  Overall survival defined as the time from the protocol therapy initiation to death from any reason
1-year and 2-year progression-free survival | 24 months
  Progression-free survival defined as the time from the protocol therapy initiation to disease progression, relapse or death from any reason.
Duration of response | 24 months
  Duration of response was defined as the time from response achievement to disease progression, relapse or death from any reason

CONTACTS AND LOCATIONS:
Overall Officials: Kirill Lepik, MD, PhD, Principal Investigator — St. Petersburg State Pavlov Medical University; Natalia Mikhailova, MD, Study Chair — St. Petersburg State Pavlov Medical University
Locations (2):
- Russia (2):
  - St. Petersburg State Pavlov Medical University, Saint Petersburg
  - N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg